CLINICAL TRIAL: NCT04882358
Title: Alfapump® DSR Feasibility Study in Subjects With Persistent Congestion Due to Heart Failure, Resistant to Loop Diuretic Treatment
Brief Title: Safety & Feasibility of DSR TherApy in Heart FAiluRe pAtients With Persistent Congestion
Acronym: SAHARA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sequana Medical N.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-CHF-006
Record Dates: First submitted 2021-04-21; First posted 2021-05-11 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Heart Failure; Volume Overload
Keywords: sodium; alfapump; direct sodium removal; diuretic resistance
MeSH Terms: conditions — Heart Failure; Edema | interventions — Drug Delivery Systems; Sodium-Glucose Transporter 2 Inhibitors; dapagliflozin

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, open label, feasibility and safety study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP 1 DIRECT SODIUM REMOVAL + SGLT-2 INHIBITOR (Experimental): SUBJECTS TREATED WITH DSR + STANDARD DOSE OF APPROVED SGLT-2 INHIBITOR
  Interventions: Device: ALFAPUMP DSR (DIRECT SODIUM REMOVAL) SYSTEM; Drug: SGLT2 inhibitor
- GROUP 2 DIRECT SODIUM REMOVAL (Experimental): SUBJECTS TREATED WITH DSR
  Interventions: Device: ALFAPUMP DSR (DIRECT SODIUM REMOVAL) SYSTEM

INTERVENTIONS:
Device: ALFAPUMP DSR (DIRECT SODIUM REMOVAL) SYSTEM — Infusion of sodium free Dextrose 10% into peritoneal cavity to remove sodium and fluid using principles of peritoneal dialysis; sodium and ultrafiltrate will be evacuated to the bladder by the alfapump
Drug: SGLT2 inhibitor — treatment with a standard dose of SGLT-2 inhibitor
  Other Names: dapagliflozin
  Arms: GROUP 1 DIRECT SODIUM REMOVAL + SGLT-2 INHIBITOR

SUMMARY:
Feasibility and safety study of the alfapump DSR system in the treatment of volume overloaded heart failure subjects receiving high doses of loop diuretics. Up to 24 subjects will be enrolled in up to 3 centres in Republic of Georgia, and randomized into 2 parallel treatment arms. Once implanted with the alfapump DSR system they will undergo DSR therapy in 2 phases: intensive treatment phase followed by maintenance treatment phase.

DETAILED DESCRIPTION:
The feasibility trial will consist of a 24-subject randomized study in volume overloaded heart failure subjects receiving high dose of loop diuretics. Subjects providing consent for participating in the clinical trial will be screened for eligibility. Once eligibility is confirmed they will be implanted with the alfapump® and a standard peritoneal infusion port. After the implant, the subject will undergo a 40 mg IV furosemide (or 1 mg IV bumetanide) diuretic challenge with timed biospecimen collection. At the start of the study treatment period, the loop diuretics treatment will be stopped. Subjects will be randomized in an unblinded fashion into one of two groups:

* Group 1 (N= 12) - treatment with a standard dose of SGLT2-inhibitor, combined with DSR treatment (PRN use of loop diuretics)
* Group 2 (N= 12) - treatment with DSR treatment (PRN use of loop diuretics) Enrolled subjects in both groups will undergo at least two weeks of intensive alfapump® DSR treatment (Phase 1) followed by a maintenance and follow-up period of 16 weeks (Phase 2).

During Phase 1 (this can be an in-patient or an out-patient setting, depending on the local standard of care practices), DSR treatment will be performed in the hospital for each subject with the baseline treatment regimen being 1L 10% dextrose (DSR infusate) with a two-hour dwell time. During this phase 1 period, there will be 2 subsequent treatment intensities: Phase 1a) Active weight reduction and Phase 1b) Weight stabilization. The active weight reduction phase (phase 1a) will start with 3 consecutive daily DSR treatment visits in all subjects. Three consecutive daily visits are required to determine the subsequent DSR treatment frequency and dose. Prior to each planned DSR treatment, the subject is evaluated (weight, vital signs, and physical exam) and blood analysis is performed. Pending this evaluation, the next DSR treatment may be held, reduced (down-titrated) or escalated (up-titration) based on the proposed titration guidelines and at the discretion of the study physician. These titration guidelines differ depending on the (sub)treatment phase(s).

Before the end of the 2 intensive weeks (phase 1), many subjects may become already euvolemic and may transition from the active weight loss phase (1a) to the weight stabilization dosing phase (1b). The transition to phase 1b is based on either the resolution of signs and symptoms of volume overload and physician opinion of euvolemia or on the worsening of creatinine by 0.5mg/dL or 1.5x the subject's baseline serum creatinine. The dosing of DSR will employ identical steps as before, but the titration guidelines are adapted in order to stabilize the weight in phase 1b (rather than continue to lose weight).

After 2 weeks of DSR (end of phase 1), the subject's condition will be evaluated via a diuretic challenge before entering the Phase 2 maintenance phase of the study. Transition to Phase 2 is recommended if all of the following criteria are met

* Clinical euvolemia is achieved (clinical assessment by investigator);
* Diuretic response during diuretic challenge is >200mmol Na or 50% increase or 50 mmol Na increase from baseline
* Stable DSR dosing was achieved If these criteria are not met, it is recommended that a 2nd 2-week Phase 1 period is utilized. To ensure ease of enrolment and compliance with the protocol, this is a recommendation rather than a protocol mandate. Up to three 2-week Phase 1 periods (6 weeks total) are allowable per protocol.

During phase 2 all subjects will receive DSR using 1L of D10 in a monthly maintenance treatment session. In case a subject exhibits weight gain greater than 2.5kg or 50% than the weight at the end of Phase 1, loop diuretics (bumetanide, chosen for its short half-life, thus minimizing the time each day the kidney is exposed to loop diuretics) may be started using a proposed dosing schedule. The maintenance phase will last 4 months after subject has started this phase 2. Total maximum study duration (screening until end of phase 2) for each subject will be 6,5 months. During the maintenance period, subjects will be followed weekly (hospital visit or telephone call). Subjects who relapse to congestion state will be undergoing additional active DSR treatment in dose and frequency as deemed required per their clinical needs by treating physician, until decongested state is reached again. In case a subject present with repeat symptoms of volume overload or decongestion, which would necessitate a repeat of phase I treatment, this will not prolong initial 4 months duration of phase 2. The recurrent decongestion will need to be reported as (S)AE and will be followed up until resolution. At the end of the phase 2 phase, each subject undergoes a diuretic challenge to evaluate diuretic response.

At the end of the phase 2 phase, subjects may elect to keep the alfapump® DSR system implanted, in agreement with the investigator. After consenting, subjects can participate in an extended follow-up with or without DSR treatments until the end of the alfapump® DSR system lifecycle (expected maximum 2 years). In other indications (not DSR) where the alfapump® is implanted, an average pump lifecycle of 10 months is observed. During the extended follow up period, no replacement of alfapump®, peritoneal access port or alfapump catheters will be performed.

The objective of the extended follow-up is to collect more long-term safety data. For subjects for whom DSR therapy appears to be offering a benefit, the investigator can elect to offer continued monthly DSR treatment at his/her discretion, in close collaboration with scientific study management team. Subjects participating in this extended follow-up will be asked to perform an additional diuretic challenge every 3 months during the extended FU to evaluate their diuretic response.

Subjects not participating in the proposed study extension as well as subjects who elected to have the alfapump® explanted at the end of the phase 2, will be proposed to participate in a minimal extended follow-up to allow investigator to contact them monthly to gather information only on loop diuretic restart and dose after the end of the study (with a maximum of 1 year after the end of phase 2 treatment period).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 years of age
2. Subject has creatinine based eGFR (MDRD or CKD-EPI formula) >30ml/min/1.73m²
3. Subject is diagnosed with heart failure including the follow-ing:

   1. nt-proBNP > 2000 pg/ml and oral diuretic dose >80mg furosemide (or >20mg torsemide or >1mg bume-tanide)
   2. at least 1 hospitalization due to HF-related volume overload within the year prior to enrolment in the study
   3. at least 2 clinical signs and symptoms of volume over-load
4. Subject has extravascular volume overload as evidenced by:

   1. Peripheral edema > trace
   2. Known fluid weight gain, or physician estimate of ≥5kg of fluid overload;
5. Subject has systolic blood pressure ≥ 100 mmHg
6. Subject is able to tolerate surgical implantation of the alfapump using local standard of care anesthesia practices

Exclusion Criteria:

1. Subject has proteinuria > 1g/l as confirmed by dipstick (≥ +++)
2. Subject presents an excessive subcutaneous fatty tissue layer at the intended location of alfapump implant, or with other characteristics which could interfere with implantation procedure or transcutaneous charging of the alfapump.
3. Subject has anemia with hemoglobin < 8g/dL
4. Subject has serum sodium < 135 mEq/L
5. Subject has clinical signs of low output heart failure
6. Subject has severe cardiac cachexia
7. Subject has history of severe hyperkalemia or screening plasma potassium > 4.5 mEq/L (K can be 4.5-5 meq/L if on 40meq or greater daily potassium supplementation and this can be stopped for the study).
8. Subject has significant non-cardiac disease or comorbidities expected to reduce life expectancy to less than 1 year.
9. Subject has cirrhosis or history of clinically significant ascites (i.e., prior large volume paracentesis) or large volume ascites on imaging or exam
10. Subject has hemodynamically significant stenotic valvular disease
11. Subject is receiving anti-coagulative or anti-platelet treatment which cannot be withheld for 5 days (replaced by bridging therapy low molecular weight heparin or unfractionated heparin) prior to and 2-3 days after alfapump DSR system implantation;
12. Subject has suffered myocardial infarction (MI), cerebro-vascular accident (CVA) or transient ischemic attack (TIA) within 90 days prior to enrolment in the study
13. Subject has history of peritonitis or history of abdominal surgery with increased risk of major abdominal adhesion as assessed by the investigator
14. Subject has any active infection or history of recurrent urinary tract infection or history of current urosepsis
15. Subject has history of renal transplant
16. Subject has history of significant bladder dysfunction expected to interfere with ability of subject to tolerate DSR pumping into bladder
17. Subject has uncontrolled diabetes with frequent hyperglycemia or Type 1 diabetes
18. Subject has urinary incontinence
19. Subject has history of type 1 diabetes, diabetic ketoacidosis, "brittle" diabetes or frequent hypoglycemia or severe hypoglycemic episodes requiring emergent intervention (ER visit or EMS response, glucagon administration or forced oral carbs) in the last 6 months
20. Subject is pregnant or is breastfeeding or intends to become pregnant during the study
21. Subject has severe peripheral artery disease
22. Subject has hypersensitivity to SGLT2 inhibitors
23. Subject is currently participating in another clinical trial
24. Subject is unable or unwilling to comply with all required study follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-05-27 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety - Treatment related SAE | up to day 156
  Rate of treatment related serious adverse events
Safety - Device related SAE | up to day 156
  Rate of Device related serious adverse events
Safety - Procedure related SAE | up to day 156
  Rate of Procedure related serious adverse events

SECONDARY OUTCOMES:
Safety - Treatment related | day 14
  Rate of treatment related serious adverse events
Safety - Treatment related | day 128
  Rate of treatment related serious adverse events
Safety - Treatment related | up to day 156
  Rate of treatment related serious adverse events
Safety - Device related | day 14
  Rate of Device related serious adverse events
Safety - Device related | day 128
  Rate of Device related serious adverse events
Safety - Device related | up to day 156
  Rate of Device related serious adverse events
Safety - Procedure related | day 14
  Rate of Procedure related serious adverse events
Safety - Procedure related | day 128
  Rate of Procedure related serious adverse events
Safety - Procedure related | up to day 156
  Rate of Procedure related serious adverse events
Safety - Device Deficiencies | day 14
  Rate of device deficiencies
Safety - Device Deficiencies | day 128
  Rate of device deficiencies
Safety - Device Deficiencies | up to day 156
  Rate of device deficiencies
Weight loss ≥ 5kgs | day 14
  % of subjects reaching weight loss of ≥ 5kgs
Weight change | day 14
  Change in weight from baseline
Weight change | day 128
  Change in weight from baseline
Weight change | up to day 156
  Change in weight from baseline

OTHER OUTCOMES:
Euvolemic state | day 14
  Time to reach euvolemic state
Euvolemic state | day 128
  Time euvolemic state is maintained in maintenance period
Restart PRN Loop diuretic treatment | up to day 156
  Time to restart of PRN loop diuretic treatment
Restart Loop diuretic treatment | up to day 156
  Time to restart of systematic loop diuretic treatment after start of DSR treatment
Time Loop diuretic treatment reaching dose | up to day 156
  Time to reach loop diuretic treatment dose ≥ loop diuretic dose prior to DSR treatment start
Time increase Loop diuretic treatment | up to day 156
  Time to loop diuretic dose increase once on therapy
Amount Loop diuretic treatment | up to day 156
  Total mg of loop diuretic administered
Change Renal function - urea | up to day 156
  Change in renal function -urea from baseline through treatment
Change Renal function - creatinin | up to day 156
  Change in renal function -creatinin from baseline through treatment
Change Hemoconcentration markers - serum hematocrit | up to day 156
  Change in hemoconcentration markers (serum hematocrit) from baseline through treatment
Change Hemoconcentration markers - serum hemoglobin | up to day 156
  Change in hemoconcentration markers (serum hemoglobin) from baseline through treatment
Hemoconcentration markers - serum albumin | up to day 156
  Change in hemoconcentration markers (serum albumin) from baseline through treatment
Change Hemoconcentration markers - total serum protein | up to day 156
  Change in hemoconcentration markers (total serum protein) from baseline through treatment
Change N-Terminal Prohormone of Brain Natriuretic Peptide (nt-ProBNP) | up to day 156
  Change in nt-proBNP from basline through treatment
Change Hemoglobin A1c | day 128
  Change in hemoglobin A1c
DSR doses | up to day 156
  Number of DSR doses per week
Amount of 10% Dextrose infusate | up to day 156
  Amount of 10% Dextrose infusate given
DSR dose adjustments | day 14
  Number of DSR dose adjustments
DSR dose adjustments | day 128
  Number of DSR dose adjustments
Sodium | up to day 156
  Net sodium loss with each DSR treatment (8 hours of DSR exposure)
Urine volume | up to day 156
  Net fluid loss with each DSR treatment (8 hours of DSR exposure)
Change 6-hour diuretic challenge response | day 14
  Change in response to 6 hour diuretic challenge from baseline
Change 6-hour diuretic challenge response | day 128
  Change in response to 6 hour diuretic challenge from baseline
Change 6-hour diuretic challenge response | up to day 156
  Change in response to 6 hour diuretic challenge from baseline
Change Plasma electrolytes - sodium | up to day 156
  Change in plasma electrolytes - Sodium from baseline
Change Plasma electrolytes - potassium | up to day 156
  Change in plasma electrolytes - potassium from baseline
Change Plasma electrolytes - magnesium | up to day 156
  Change in plasma electrolytes - magnesium from baseline
Change Plasma electrolytes - calcium | up to day 156
  Change in plasma electrolytes - calcium from baseline
Change Plasma electrolytes - phosphor | up to day 156
  Change in plasma electrolytes - phosphor from baseline
DSR dwell time | up to day 156
  Dwell time per DSR treatment
Change Bio-impedance vector analysis | up to day 156
  Change in Bio-impedance vector analysis
Ultrafiltration | up to day 156
  Total ultrafiltration
Volume | up to day 156
  Total volume removed
Glucose | up to day 156
  Total glucose resorption during DSR treatment

CONTACTS AND LOCATIONS:
Overall Officials: TAMAZ SHABURISHVILI, MD, Principal Investigator — TBILISI HEART & VASCULAR CLINIC
Locations (2):
- Georgia (2):
  - Israeli-Georgian Medical Research Clinic Helsicore, Tbilisi
  - Tbilisi Heart & Vascular Clinic, Tbilisi

IPD SHARING:
Plan to Share IPD: No
No IPD data will be shared with other researchers

REFERENCES:
- [Derived] Rao VS, Ivey-Miranda JB, Cox ZL, Moreno-Villagomez J, Ramos-Mastache D, Neville D, Balkcom N, Asher JL, Bellumkonda L, Bigvava T, Shaburishvili T, Bartunek J, Wilson FP, Finkelstein F, Maulion C, Turner JM, Testani JM. Serial direct sodium removal in patients with heart failure and diuretic resistance. Eur J Heart Fail. 2024 May;26(5):1215-1230. doi: 10.1002/ejhf.3196. Epub 2024 Mar 31. PMID 38556717